CLINICAL TRIAL: NCT02412267
Title: An Open-label, Non-randomized Phase 2 Study of Ofatumomab (O) in Combination With ICE (Ifosfamide, Carboplatin, Etoposide)-Chemotherapy in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of Ofatumomab in Combination With ICE-chemotherapy in Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: DLBL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1001
Record Dates: First submitted 2015-03-31; First posted 2015-04-09 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ofatumumab; Ifosfamide; Carboplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- O-ICE (Experimental): O-ICE:
  Ofatumumab 1000mg intravenous (IV) infusion on Day 1 and Day 8 of cycle 1 of the salvage chemotherapy, and thereafter on Day 1 of each cycle; Ifosfamide 1667 mg/m2 IV infusion over 2 hours on days 1,2,3 of each cycle; Carboplatin 5 x ((25 + Creatinine clearance (CrCl)) IV in 250 ml Normal Saline over 1 hour on day 1 of each cycle; Etoposide 100mg/m2/day IV infusion day 1,2,3 over 45 to 60 minutes of each cycle.
  Interventions: Drug: O-ICE (ofatumumab, Ifosfamide, Carboplatin, Etoposide)

INTERVENTIONS:
Drug: O-ICE (ofatumumab, Ifosfamide, Carboplatin, Etoposide) — Ofatumab in combination with ICE (Ifosfamide, Carboplatin, Etoposide) are given to subjects according to protocol schedule
  Other Names: Arzerra, Mitoxana, Paraplatin, Etopophos

SUMMARY:
The purpose of this study is to determine the efficacy and safety of ofatumomab in combination with ICE chemotherapy in subjects with relapsed/refractory DLBCL following failure to combination rituximab and anthracycline based chemotherapy. Participants with the option of potentially curative stem cell therapy may proceed to high dose chemotherapy and stem cell rescue. Participants with disease not considered curable with stem cell therapy, ineligible for or decline stem cell therapy may receive up to a maximum of 6 cycles of study drugs.

DETAILED DESCRIPTION:
This is a Phase II, single-arm, non randomized, safety and efficacy study of ofatumumab in combination with salvage ICE chemotherapy (O-ICE) in 61 subjects with relapsed or refractory aggressive B cell lymphoma.

O-ICE would be administered as an inpatient. The cycles are administered at 3 weeks intervals for ICE.

Study subjects who are candidates for high dose chemotherapy (HDC) and autologous stem cell rescue (ASCR) would receive one or two more cycle of ICE salvage chemotherapy with ofatumumab before stem cell mobilization. G-CSF at 10 ug/kg per day after the third or forth cycle of treatment (at the discretion of the treating physician) would be administered until the end of leukapheresis for stem cell mobilization. After the third or forth cycle of salvage chemotherapy, leukapheresis was initiated until a collection of more than 5 x 106 CD34 cells/kg white blood or 5 procedures were performed, whichever occurred first. Collection of <2x106 CD34+ cells/kg from peripheral blood will be considered mobilization failure for the purposes of the study. Leukapheresis and cryopreservation will be performed according to hospital practice. High dose chemotherapy will be administered as per our institution's protocol.

Study subjects who are not candidates for HDC and ASCR would receive at most 6 cycles of salvage chemotherapy with ofatumumab.

Subjects who progressed on treatment would be taken off study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory or relapsed CD20 positive DLBCL following rituximab combined with chemotherapy.
2. Participants must have measurable disease
3. ECOG performance status 0-2
4. Unless due to lymphomatous involvement, participants must have adequate organ and marrow function as defined below:

   * Hemoglobin ≥ 10g/dL
   * Absolute neutrophil count ≥ 1500/mm3
   * Platelets ≥ 100 000/mm3
   * ALT and AST ≤ 3 x upper limit of normal (ULN),
   * Total serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
5. Fully recovered (≤ Grade 1 or returned to baseline or deemed irreversible) from the acute effects of prior cancer therapy before initiation of study drug
6. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Any previous cancer therapy for lymphoma, with the exception of Rituximab in combination with chemotherapy (not more than 1 prior line of chemotherapy)
2. Participants who have had systemic anti-cancer therapy within 3 weeks (8 weeks for nitrosoureas or mitomycin C) prior to study entry
3. Participants who have had radiotherapy and/ or major surgery within 3 weeks prior to study entry
4. Participants who have had systemic corticosteroids for the purpose of treating lymphoma within 2 weeks prior to study entry are ineligible. Patients receiving stable (not increased within the last month) chronic doses of systemic corticosteroids with a maximum dose of 20 mg of prednisolone (or equivalent) per day are eligible if they are being given for disorders other than lymphoma
5. Concurrent use of any other anti-cancer therapies or study agents.
6. Presence of symptomatic or uncontrolled brain or central nervous system lymphomatous lesions
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant cardiac disease including a history of cardiac disease or congestive heart failure > NYHA class 2, unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months, significant cardiac arrhythmias and/ or requiring anti-arrhythmics; pulmonary disease; liver diseases such as cirrhosis, chronic active or persistent hepatitis; or acute/ chronic medical/ psychiatric illness/ social situations or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or limit compliance with study requirements, or interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
8. Known or suspected hypersensitivity to study treatments.
9. History of HIV or Hepatitis C
10. Individuals with a history of a different malignancy, other than treated cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR other primary malignancy is neither currently clinically significant nor requiring active intervention.
11. Pregnant or lactating women.
12. Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of ofatumumab therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence. Women of childbearing potential must have a negative pregnancy test prior at screening.
13. Male subjects unable or unwilling to use adequate contraception methods from the time of first dose of study medication until one year after the last dose of ofatumumab.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by the new international criteria proposed by Cheason for response in non Hodgkin's lymphoma at the end of cycle 2 ofatumomab | 5 years
  Response (partial or complete response) status will be evaluated following two cycles of ofatumumab in combination with ICE chemotherapy

SECONDARY OUTCOMES:
Progression free survival as measured from time of treatment start to time of disease progression | 5 years
  Progression evaluation will follow the new international criteria proposed by Cheason for response in non Hodgkin's lymphoma
Safety and tolerability of Ofatumomab in combination with ICE chemotherapy as measured by CTCAE | 5 years
  Adverse events will be graded following CTCAE (Common Terminology Criteria for Adverse Events) V4.03, and the relationship to the study treatment will be assessed by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Soon Thye Lim, Dr, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore